CLINICAL TRIAL: NCT05863832
Title: Single Center, Open Label, Controlled Study to Assess the Safety & Efficacy of Oral Ciprodiazole Versus Currently Used Ciprofloxacin & Metronidazole Tablets in Pelvi-abdominal Infections and Following IV Antibiotics in Post-operative Period
Brief Title: Study to Assess the Safety & Efficacy of Oral Ciprodiazole Versus Currently Used Ciprofloxacin & Metronidazole
Acronym: CIPRO-001
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MinaPharm Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIPRO-001
Record Dates: First submitted 2023-04-06; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-04

CONDITIONS: Surgical Site Infections
MeSH Terms: conditions — Surgical Wound Infection | interventions — Ciprofloxacin; Metronidazole

STUDY DESIGN:
Intervention Model Description: They will be randomized by computer, into 2 treatment groups; Ciprodiazole ® tablets (Ciprofloxacin/Metronidazole) versus currently used Ciprofloxacin Tablets & Metronidazole tablets
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprodiazole (Experimental): Ciprodiazole Tablets: (Ciprofloxacin 500 mg & Metronidazole 500 mg), 1 tablet every 12 hours up to 15 days
  Interventions: Drug: Ciprodiazole
- Ciprofloxacin 500 mg Tablets & Metronidazole 500 mg tablets (Active Comparator): Ciprofloxacin 500 mg Tablets: 1 tablet every 12 hours up to 15 days
  Metronidazole 500 mg tablets: 1 tablet every 8 hours up to 10 days
  Interventions: Drug: Ciprofloxacin Tablets & Metronidazole tablets

INTERVENTIONS:
Drug: Ciprodiazole — Ciprofolxacin 500 mg / Metronidazole 500 mg
  Arms: Ciprodiazole
Drug: Ciprofloxacin Tablets & Metronidazole tablets — Ciprofolxacin 500 mg + Metronidazole 500 mg
  Arms: Ciprofloxacin 500 mg Tablets & Metronidazole 500 mg tablets

SUMMARY:
This study aims to assess the safety & efficacy of Oral Ciprodiazole® versus currently used Ciprofloxacin Tablets & Metronidazole tablets in pelvi-abdominal infections and following IV antibiotics in post-operative period, for pelvi-abdominal surgeries or acute conditions

DETAILED DESCRIPTION:
Primary Objective

1. Primary Safety:

   To compare safety of oral Ciprodiazole ® tablets (Ciprofloxacin/Metronidazole) versus currently used Ciprofloxacin Tablets & Metronidazole tablets for pelvi-abdominal infections, either non-operative or post-operative following IV antibiotics.
2. Primary Efficacy:

To compare efficacy of oral Ciprodiazole ® tablets (Ciprofolxacin/Metronidazole) versus currently used Ciprofloxacin Tablets & Metronidazole tablets for pelvi-abdominal infections, either non-operative or post-operative following IV antibiotics.

Secondary Objective

1. Secondary Safety:

   * Presence of any signs/symptoms of post-operative wound infection such as redness, fever or wound discharge.
   * Presence of undesirable effects on total leukocyte count and liver enzymes (SGOT& SGPT)
2. Secondary Efficacy:

   * To compare the complete resolution or improvement of Pelvi-abdominal infection between ciprodiazole® versus combined treatment, based on pelvi-abdominal ultrasound and others
   * To compare the days for complete healing of post-operative wounds between ciprodiazole® versus combined treatment

STUDY DURATION:

* Subjects will be enrolled for 12 months including screening visit
* Follow up for 15 days from enrolment

STUDY POPULATION:

312 Egyptian Patients with pelvi-abdominal infection or started IV antibiotics in post-operative period, for pelvi - abdominal surgeries and/or acute conditions

ASSESSMENT SCHEDULE:

Subjects will be enrolled for 12 months including screening visit

* Visit 1: Screening and treatment initiation visit, Day 0
* Follow-up 1 visit: Day 8 (+/-) 3 days
* Follow-up 2 visit & End of study visit: Day 15 (+/-) 3 days

ELIGIBILITY:
Inclusion Criteria:

1. Egyptian male and female patients aged between 18-65 years' old
2. Subjects having pelvi-abdominal infections such as and not limited to: Ulcerative Colitis, Diverticulitis, Cholecystitis and Pelvic Inflammatory Diseases (PID), as oophoritis and salpingo-oophoritis.
3. Subjects during post-operative period for pelvi-abdominal surgery and following IV medication with Metronidazole injection plus third generation cephalosporin.
4. Subjects who are willing to sign Informed Consent Form (ICF) and ready to comply with the protocol for the duration of the study

Exclusion Criteria:

1. Subjects with a history of hypersensitivity to any of the active ingredients of the treatments used
2. Subjects who are receiving or received any other antibiotics during the previous two weeks, rather than IV treatment in the first post-operative 48 hours, mentioned in the protocol
3. Subjects with Pelvi-abdominal infection and performed surgery after failure of oral antibiotics.
4. Subjects having surgeries such as colorectal surgeries.
5. Subjects with any medical condition requiring the usage of the following medications:

   * Drugs that induce microsomal liver enzymes, such as Phenytoin or Phenobarbital.
   * Drugs that decrease microsomal liver enzymes activity, such as cetrimide.
   * Theophylline
   * Corticosteroids
   * Antacids containing magnesium and aluminum, supplements and other products containing calcium, iron or zinc
   * Tizanidine
6. Subjects with uncontrolled diabetes mellitus; FBG > 200 mg/ml
7. All subjects with renal impairment (S. Creatinine > 1.5 mg/dL)
8. All subjects with hepatic impairment (Child-Pugh Score B-C)
9. Subjects with liver enzymes (SGOT & SGPT > 2 Normal range)
10. Pregnant or breast-feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Up to 15 Days
  Incidence of serious/ non-serious adverse events
Wounds healing | Up to 15 Days
  Complete healing of the of post-operative wounds
Resolution of pelvi-abdominal infection | Up to 15 Days
  Complete resolution for pelvi-abdominal infection, based on clinical response and/or pelvi-abdominal ultrasound and others

SECONDARY OUTCOMES:
Signs of post-operative wound infection | Up to 15 Days
  Presence of any signs of post-operative wound infection such as redness, fever or wound discharge
Change in Safety Lab measures | Up to 15 Days
  Change in Total Leukocyte count and serum Liver enzymes (SGOT, SGPT) between baseline (visit 1) to End of study visit (Follow up 2 V)
Infection outcome | Up to 15 Days
  Complete resolution, improvement, failure or relapse of pelvi-abdominal infection, based on pelvi-abdominal ultrasound and/or clinical response
Healing Days | Up to 15 Days
  Days for complete healing of post-operative wounds between the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Dr El Kased, PhD, Principal Investigator — Faculty of Medicine - Menoufia University
Locations (1):
- Faculty of Medicine - Menofia University, Shibīn al Kawm, Menofia, Egypt

DOCUMENTS (3):
  • Study Protocol (2022-03-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT05863832/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT05863832/SAP_001.pdf
  • Informed Consent Form (2022-03-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT05863832/ICF_002.pdf